CLINICAL TRIAL: NCT00296387
Title: Comparison of the Effects Noted in The ApoB/ApoA-I Ratio Using Rosuvastatin and Atorvastatin in Patients With acUte Coronary Syndrome - CENTAURUS
Brief Title: Effects in The ApoB/ApoA-I Ratio Using Rosuvastatin and Atorvastatin in Patients With Acute Coronary Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D3560L00052; CENTAURUS
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2007-12-17 (Estimated); Status verified 2007-12

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Rosuvastatin Calcium; Atorvastatin

INTERVENTIONS:
Drug: Rosuvastatin
Drug: Atorvastatin

SUMMARY:
The purpose of this study is to see if rosuvastatin compared to Atorvastatin is effective in treating ACS by decreasing the ApoB/ApoA-1 ratio and if starting statin within 24 h following the onset of the first symptoms is beneficial compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Hospital admission for ACS with chest pain or discomfort occurring during rest or with minimal exertion,
* Percutaneous coronary intervention (PCI) planned,
* Evidence of coronary artery disease

Exclusion Criteria:

* Hypersensitivity to statins
* Any cholesterol lowering medication taken within 1 month prior V1
* Sustained ST-segment elevation on ECG

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1160 (Estimated)
Dates: Start 2006-01; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Percentage changes in ApoB/ApoA-I levels | from Day 0 to 3 months

SECONDARY OUTCOMES:
Percentage changes in LDL-C | from Day 0 to 1 month and 3 months
Percentage changes in the hs-CRP and AUC of hs-CRP levels | from Day -6 to Day 0
Percentage changes in ApoA-I | from Day 0 to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca France Medical Director, MD, Study Director — AstraZeneca
Locations (102):
- Belgium (9):
  - Research Site, Aalst
  - Research Site, Bonheiden
  - Research Site, Bouge
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Hasselt
  - Research Site, Huy
  - Research Site, La Louvière
  - Research Site, Leuven
- Canada (17):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Saint John, New Brunswick
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Regina, Saskatchewan
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- France (34):
  - Research Site, Amiens
  - Research Site, Annecy
  - Research Site, Arras
  - Research Site, Avignon
  - Research Site, Boulogne-Billancourt
  - Research Site, Caen
  - Research Site, Cholet
  - Research Site, Créteil
  - Research Site, Dijon
  - Research Site, Eaubonne
  - Research Site, Évecquemont
  - Research Site, Falaise
  - Research Site, La Roche-sur-Yon
  - Research Site, Lagny-sur-Marne
  - Research Site, Le Coudray
  - Research Site, Le Mans
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Metz
  - Research Site, Montpellier
  - Research Site, Nevers
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, Pessac
  - Research Site, Reims
  - Research Site, Rouen
  - Research Site, Saint-Herblain
  - Research Site, Suresnes
  - Research Site, Toulouse
  - Research Site, Tourcoing
  - Research Site, Tours
  - Research Site, Valenciennes
  - Research Site, Vannes
  - Research Site, Villeurbanne
- Research Site, Athens, Greece
- Hungary (4):
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Pécs
  - Research Site, Zalaegerszeg
- Ireland (3):
  - Research Site, Dublin
  - Research Site, Galway
  - Research Site, Limerick
- Italy (13):
  - Research Site, Bari, Apulia
  - Research site, Cosenza, Basilicate
  - Research Site, Benevento, Campania
  - Research Site, Mantova, Lombardy
  - Research Site, Rozzano (Milano), Lombardy
  - Research Site, Catania, Sicily
  - Research Site, Pisa, Tuscany
  - Research Site, Perugia, Umbria
  - Research Site, Verona, Veneto
  - Research Site, Bolzano
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Roma
- Portugal (7):
  - Research Site, Aveiro
  - Research Site, Braga
  - Research Site, Carnaxide
  - Research Site, Faro
  - Research Site, Funchal
  - Research Site, Leiria
  - Research Site, Vila Real
- Spain (8):
  - Research Site, Zaragoza, Aragon
  - Research Site, Toledo, Castille-La Mancha
  - Research Site, Tarragona, Catalonia
  - Research Site, Fuenlabrada(Madrid), Madrid
  - Research site, Madrid, Madrid
  - Research Site, Vigo, Pontevedra
  - Research Site, Sant Joan d'Alacant, Valencia
  - Research Site, Seville
- Tunisia (4):
  - Research Site, BAB Saâdoun Tunis
  - Research Site, SIDI Daoud Tunis
  - Research Site, Sousse
  - Research Site, Tunis

REFERENCES:
- [Derived] Lablanche JM, Leone A, Merkely B, Morais J, Alonso J, Santini M, Eha J, Demil N, Licour M, Tardif JC; CENTAURUS investigators. Comparison of the efficacy of rosuvastatin versus atorvastatin in reducing apolipoprotein B/apolipoprotein A-1 ratio in patients with acute coronary syndrome: results of the CENTAURUS study. Arch Cardiovasc Dis. 2010 Mar;103(3):160-9. doi: 10.1016/j.acvd.2010.01.005. Epub 2010 Apr 8. PMID 20417447